CLINICAL TRIAL: NCT07258381
Title: A Multicenter, Randomized Controlled Trial on the Efficacy of Mailuo Shutong Pills in Treating Diabetic Wounds With Damp-Heat Toxin Accumulation Syndrome
Brief Title: Mailuo Shutong Pills for Diabetic Wound Healing: A Multicenter Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Head of Wound Healing Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2025-DW-ChineseMed：MLST
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Wound; Chronic Wound Care
Keywords: diabetic wound; chronic wound care

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Based on the clinical standard treatment plan, oral administration of Maoluo Shutong Pills was administered for 2 weeks
  Interventions: Drug: Mailuo Shutong Pills
- Control group (Sham Comparator): the clinical standard treatment plan
  Interventions: Drug: Blank control

INTERVENTIONS:
Drug: Mailuo Shutong Pills — a medicine that treating Diabetic Wounds with Damp-Heat Toxin Accumulation Syndrome
  Arms: Experimental group
Drug: Blank control — Blank control
  Arms: Control group

SUMMARY:
Mailuo Shutong Pills are a Chinese patent medicine approved for market release by the China Food and Drug Administration (CFDA) in 2009. It is formulated by integrating five classical herbal formulas, including Ermiao San, Simiao Yongan Tang, and Zhijing San. Its composition is as follows: Honeysuckle Flower (Jinyinhua) serves as the principal component (Jun herb) for clearing heat and detoxifying; Astragalus Root (Huangqi) for tonifying qi, expelling toxin, and promoting diuresis; Phellodendron Bark (Huangbai), Atractylodes Rhizome (Cangzhu), and Coix Seed (Yiyiren) act as deputy components (Chen herbs) to clear heat and resolve dampness; Chinese Angelica (Danggui), Peony Root (Baishao), and Licorice Root (Gancao) alleviate spasm and pain; Figwort Root (Xuanshen) cools the blood, clears heat, drains fire, detoxifies, and softens hard masses. Leeches (Shuizhi), Centipede (Wugong), and Scorpion (Quanxie) serve as assistant components (Zuo herbs) to invigorate blood, resolve stasis, attack toxicity, dissipate nodules, and unblock collaterals to relieve pain. Licorice Root (Gancao) also harmonizes the various components in the formula as the envoy component (Shi herb). The complete formula possesses the effects of clearing heat and detoxifying, dissolving stasis and unblocking collaterals, and dispelling dampness and reducing swelling. It is indicated for various conditions differentiated in Traditional Chinese Medicine (TCM) as presenting with a pattern of dampness-heat and stasis obstruction, such as superficial thrombophlebitis and deep vein thrombosis in the non-acute stage.

Some studies suggest that Mailuo Shutong Pills may have a positive effect in the field of wound healing, for example, by significantly reducing the release of inflammatory mediators such as IL-1β, IL-6, CRP, and TNF-α caused by inflammatory diseases [11-13], and accelerating the healing of diabetic foot wounds [14]. Clinical guidelines, including the "Clinical Application Guide for Chinese Patent Medicines - Diabetes Volume" from the Diabetes Branch of the China Association of Chinese Medicine and the "Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment Guidelines for Diabetic Foot" from the Chinese Medical Doctor Association, recommend Mailuo Shutong Pills for the treatment of diabetic foot ulcers [15]. However, the current related evidence-based medical evidence is insufficient. We have also observed that the adjunctive use of Mailuo Shutong Pills does not guarantee a shortened healing time for all patients with diabetic wounds. From a TCM perspective, the presence of a dampness-heat and stasis obstruction pattern is a key factor determining the efficacy of adjunctive Mailuo Shutong therapy. For Western medicine practitioners, tongue diagnosis presents a practicable factor for assessing pattern manifestation. Therefore, based on differences in patient patterns and using tongue appearance as an inclusion/exclusion criterion, to screen for the indications of Mailuo Shutong Pills combined with existing standard treatment for diabetic wounds constitutes an effective technical approach to address the aforementioned issues.

Consequently, this study aims to explore the indications for Mailuo Shutong Pills in diabetic wounds and obtain evidence-based medical evidence for its clinical efficacy within an integrated Chinese-Western medicine approach. Furthermore, to enhance the study's external validity and participant recruitment efficiency, thereby accelerating the research progress, this study is designed as an exploratory trial conducted across multiple centers.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of type 1 or type 2 diabetes mellitus;
* the type of wound is an ulcer, with an ulcer area ranging from 1 to 40cm ²;
* the wound etiology is diabetic, mainly abnormalities in blood glucose, resulting in poor or prolonged healing and requiring standard wound therapy;
* The traditional Chinese medicine diagnosis is Damp-Heat Toxin Accumulation Syndrome;
* voluntary participation in the study and signing of an informed consent form.

Exclusion Criteria:

* Diagnosis of a Cold Pattern according to Traditional Chinese Medicine (TCM) differentiation, manifested as: pale, enlarged, and tender tongue with a white, moist or glossy coating; pallor; pale lips; aversion to cold with a preference for warmth; and loose stools.
* Pregnancy or lactation.
* Presence of severe, uncorrected systemic diseases, such as acute myocardial infarction, heart failure, hepatitis, shock, or respiratory failure.

Active bleeding within the wound that prevents the implementation of standard wound care.

* Severe laboratory abnormalities: serum albumin < 20 g/L; hemoglobin < 60 g/L; or platelet count < 50 × 10⁹/L.
* Diagnosis of advanced malignant tumor.
* Active phase of an autoimmune disease.
* History of hypersensitivity to Mailuo Shutong Pills or Mailuo Shutong Granules.
* Inability to cooperate with the study procedures or presence of psychiatric disorders.
* Any other condition considered by the investigator as a clear, unmodifiable factor adversely affecting wound healing, making the candidate unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
wound area reduction rate | Day14 ± 2
  Pre-treatment area minus post-treatment area, then divided by pre-treatment area

SECONDARY OUTCOMES:
wound healing rate | Day14 ± 2
  Percentage of healed wounds to total cases by D14
Granulation tissue status | Day 0/Day 14 ± 2
  They were classified as healthy granulation, inflammatory granulation, infected granulation, oedematous granulation, and aged granulation. D0/D14, wound granulation tissue status was recorded separately
wound infection control | Day 0/Day 14 ± 2
  0 points for no infection, 1 point for reduction of localised infection; 2 points for maintenance or exacerbation of localised infection; 3 points for disseminated infection; record D0/D14, the status of the wound infection and record the scoring results respectively
Tongue appearance | Day 0, Day 7±2 and Day 14±2
  According to the tongue image photography SOP, record the tongue images

IPD SHARING:
Plan to Share IPD: Undecided